CLINICAL TRIAL: NCT04164771
Title: Effect of Aerobic Training and Moringa Oleifera on Dyslipidemia and Cardiac Endurance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Muhammad Safdar Ali (Unknown)
Responsible Party: Principal Investigator, NASEER AHMED, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NA 125
Record Dates: First submitted 2019-11-07; First posted 2019-11-15 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Dyslipidemias
Keywords: Aerobic training; Moringa; Cardioprotection
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moringa Group (Experimental): Participants will receive 5-7g of moringa diet daily for 6 weeks.
  Interventions: Other: Aerobic training and Moringa Oleifera
- Aerobic training Group (Experimental): Participants will receive 5-7g of moringa diet daily and will do 30 minutes of aerobic training daily for 6 weeks.
  Interventions: Other: Aerobic training and Moringa Oleifera
- Moringa and Aerobic training (Experimental): Participants will do 30 minutes of aerobic training daily for 6 weeks
  Interventions: Other: Aerobic training and Moringa Oleifera
- Control Group (T4) (No Intervention): Participants will not recieve any treatment

INTERVENTIONS:
Other: Aerobic training and Moringa Oleifera — Aerobic exercises/training refers to any type of rhythmic, continuous physical activities that use large group of muscles like walking, running, cycling, and swimming consuming additional amount of energy while Moringa Oleifera a plant from the family Moringacea, its products are used as a health supplement introduced in Africa and south Asian countries to cure many diseases and improve health status
  Arms: Aerobic training Group; Moringa Group; Moringa and Aerobic training

SUMMARY:
Aerobic training is essential for maintaining and improving physical performance and has a positive effect on physiological functions as well as anthropometric characteristics. It also has positive effect on cardiovascular health and carries a number of beneficial effects on the whole body functions and systems. Aerobic training can also decrease the risk of heart disease in the individual's life.The Moringa leaves are the rich source of minerals, vitamins and other essential phytochemicals. Moringa leave have found to be very effective in many disease particularly diabetic, blood pressure, dyslipidemia and cancer.

DETAILED DESCRIPTION:
Aerobic training is an important component for health in daily life as well as sports performance. Aerobic training improves overall health, reduces body fat, maintain body weight, resting blood pressure (systolic and diastolic), maximal oxygen consumption adequate blood supply and provision of oxygen to the body muscles .The studies reveal that aerobic training is valuable for improving cardiovascular health, fitness and quality of life. On account of lack of aerobic engagement around 17 % of the population suffer from heart related ailment, 12 % from diabetes and 10 % from breast cancer. American College of Sports Medicine suggested that 30 minutes of aerobic workout has progressive effects on physical fitness and especially on chronic diseases. Physically fit individuals have got the potential to affectively cope with stress and anxiety and coronary arteries diseases. Aerobic training can raise maximal oxygen uptake, which means body adapts to use oxygen more efficiently during physical activities. Resultantly, the heart becomes efficient and stronger; meaning that the heart doesn't have to work hard to pump blood in resting position. Aerobic training decreases resting heart rate and may increase blood volume and blood plasma. Moringa Oleifera a plant from the family Moringacea, its products are used as a health supplement introduced in Africa and south Asian countries to cure many diseases and improve health status . Moringa leaves are rich source of vitamins and protein. The Moringa oleifera leaves, flowers, seeds and pods are commonly used as vegetables diet in different regions of south Asia. Moringa plant products are sources of vitamin A, b, C and proteins, including the essential amino acids. Moringa Oleifera leaves can be merged in the feed of birds, animals and human which provide wonderful source of protein other than expensive ingredients. The Moringa oil is used in cooking products as well as for lubrication. There are scientific indications that Moringa Oleifera holds therapeutic potential for hyperlipidemia, diabetes and cardiovascular diseases. The use of herbal supplements has increased rapidly during the first decade of the twentieth century. The nutrients of Moringa are considered to be useful for disorders including skin disease, malnutrition and sexual problem.Different experimental studies has described that Moringa oleifera leaves have therapeutic potential for chronic hyperglycemia and dyslipidemia . Moringa Oleifera is used as a hypolipidemic medication to improve the lipid profile of rats fed on atherogenic diet. Moringa Oleifera intake is more effective in prevention than in treatment of hyperlipidemia.It is documented that overuse of Moringa supplements can cause high increase of iron. Hence, a daily 70 g quantity of Moringa is recommended to be batter and preventive for accumulation of nutrients.This research study is due to be conducted to determine the effect of aerobic training and Moringa Oleifera on dyslipidemia and cardiac endurance

ELIGIBILITY:
Inclusion Criteria:

* Healthy and no medical conditions.
* LDL level should be 160-189 mg/dl
* HDL level should be < 40 mg/dl
* Tri glyceride level should be 200-499 mg/dl
* Total cholesterol level should be > 200 mg/dl).
* Beep Test score should be less than 10.5 or less than 40% vo2 max

Exclusion Criteria:

* Any disease condition as anemia, physical injuries, chronic disease
* Not capable of doing aerobic training

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Positive effect of aerobic training and Moringa Oleifera on dyslipidemia and cardiac endurance | 6 weeks
  Change in level of HDL, LDL and triglyceride, impact on cardiac endurance

CONTACTS AND LOCATIONS:
Overall Officials: Naseer Ahmed, Ph.D, Principal Investigator — Agha Khan Hospital

IPD SHARING:
Plan to Share IPD: No